CLINICAL TRIAL: NCT06768099
Title: Reducing Disparities for Children in Rural Emergency Resuscitation (RESCU-ER): Developing and Testing the Acceptability and Feasibility of an Integrated Linear Cognitive Aid for Pediatric Resuscitation in a Pilot RCT
Brief Title: A Clinical Trial to Study the Feasibility and Acceptability of an App to Support Pediatric Resuscitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeanne-Marie Guise, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023P000386; R01HL141429 (NIH)
Record Dates: First submitted 2024-12-30; First posted 2025-01-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Emergency Medicine; Resuscitation; Pediatrics; Emergency Medical Services; Arrest Cardio Respiratory
Keywords: Pediatric emergency medical services; Rural-urban health disparities; Child mortality; Adverse safety events (ASEs); Prehospital pediatric care; Cognitive aid; Randomized controlled trial (RCT); Emergency resuscitation; Out of hospital Cardiac arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: We propose to conduct a pilot feasibility randomized control trial of a mobile app that provides AHA cardiac resuscitation guidance. We will perform high-fidelity simulation of two children's resuscitation scenarios. Teams will be randomized to: 1) perform both resuscitations with their current standard with existing cognitive aids or 2) perform both resuscitations using our mobile app. The order of the scenarios will be randomized for each team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Current Standard with Existing Cognitive Aids (No Intervention): We will perform in situ high-fidelity simulation of two critical children's emergency resuscitation scenarios using the current standard of care with existing cognitive aids.
- Linear Cognitive Aid (Experimental): We will perform in situ high-fidelity simulation of two critical children's emergency resuscitation scenarios using a linear cognitive aid
  Interventions: Other: Linear Cognitive Aid

INTERVENTIONS:
Other: Linear Cognitive Aid — Key features of this tool include:
  * Minimal input: Teams input the patient's age and clinical scenario (e.g. arrest, childbirth, or trauma).
  * Linear logic: Based on initial simple input, the tool provides straightforward guidance without requiring multiple Y/N input or advanced decision-making.
  * Guidance based on individual characteristics: The tool tailors AHA guidance for the specific emergency scenario to the individual patient's size (estimated by age), emphasizing key interventions for the individual scenario and giving appropriate size-based guidance regarding choice of equipment, medication dosage, and resuscitation technique (e.g., chest compression depth).
  * Time-based and on-demand guidance: Based on the time elapsed from the start of the resuscitation, the app will provide audio guidance regarding the next key steps.
  Arms: Linear Cognitive Aid

SUMMARY:
The goal of this clinicial trial is to test the acceptability and feasibility of linear cognitive aid intervention to support EMS teams in responding to pediatric emergencies. We are testing the hypothesis that cognitive aids with linear logic will be feasible to use and acceptable to EMS teams in urban and rural areas.

Researchers will compare technical performance, teamwork, and self-assessed cognitive load of participants to see the difference between performing resuscitations using their current standard with existing cognitive aids and using our linear cognitive aid.

Participants' teams will:

* perform in situ high-fidelity simulation of two critical children's resuscitation scenarios
* be randomized to 1) perform both resuscitations with their current standard with existing cognitive aids or 2) perform both resuscitations using our linear cognitive aid.

ELIGIBILITY:
Inclusion Criteria:

* Active public, private, volunteer, hospital-based, or third-party EMS providers
* Speaks and understands English
* Age 18 and over

Exclusion Criteria:

- Not clinically active

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to Achieve AHA Technical Milestones | 10 minute simulation
  Time stamps for achieving completion of clinically recommended steps according to AHA guidance in minutes and seconds over a total 10 min simulation session. Less time taken is better performance.

SECONDARY OUTCOMES:
Teamwork | Cumulative evaluation over each 10 minute simulation
  Teamwork will be evaluated in real time using the validated Clinical Teamwork Scale (CTS™) over each 10 minute simulation. The scale ranges from 0 to 10, with 0 being "unacceptable" and 10 being "perfect."
Cognitive load | Cumulative evaluation over each 10 minute simulation
  Cognitive load will be self-assessed after each 10 minute simulation, using the NASA-TLX, a previously validated and widely used tool that measures mental, physical, and temporal demand, overall performance, effort, and frustration level to create an overall task load index for each team member. The scale has a range of 0 to 100 with a higher score indicating higher cognitive load.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - 20 Overland 4th floor, Boston, Massachusetts
  - BIDMC, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
This study does not involve patients. It involves prooviders responding to simulated emergencies and is part of quality and safety and is protected under this.

REFERENCES:
- [Derived] Lee SA, Trujillo D, Meckler GD, Eriksson C, Huynh T, Bahr N, Sanjeevi J, Hansen M, Guise JM. RESCUER mobile app to support pediatric resuscitation: Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2025 Oct 8;48:101558. doi: 10.1016/j.conctc.2025.101558. eCollection 2025 Dec. PMID 41142041